CLINICAL TRIAL: NCT01888926
Title: Investigating the Plastic Effects of Repetitive Paired Associative Stimulation (rPAS) in Dystonia
Brief Title: The Effects of Repetitive Paired Associative Stimulation in Dystonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130163; 13-N-0163
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2016-08-02

CONDITIONS: Dystonia
Keywords: rPAS; Dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- People with dystonia have serious muscle contractions that cause abnormal movements or postures. This significantly affects their daily lives. The common type is called organic. The other type is psychogenic. People with this type have typical symptoms plus some psychological effects. Researchers will look at how rapid transcranial magnetic stimulation (rTMS) of the brain combined with stimulation of a nerve affects the ability to detect sensations. They will compare the responses of people with different types of dystonia. They will also compare the responses of people with dystonia to responses of people without it. This study may help us learn more about the nature of different types of dystonia.

Objectives:

- To see whether TMS combined with nerve stimulation affects the brain differently in people with different types of dystonia and those without dystonia.

Eligibility:

* Individuals at least 18 years old, who are right-handed and have dystonia.
* Healthy volunteers at least 18 years old.

Design:

* Participants will have two clinical visits. Each visit will be a few hours long. They can be done on the same day.
* Participants will be screened with a medical history and physical exam.
* Participants will take several sensory tests. For these tests, electrodes will be placed on their skin. The participants will feel small electric shocks during some of the tests.
* Participants will undergo TMS. For 2 minutes, quick electrical currents will pass through a wire coil placed on their head. As this happens, researchers will ask the participants to move certain muscles.

DETAILED DESCRIPTION:
Objective:

To investigate the effects of pairing brain and peripheral nerve stimulation in organic and psychogenic dystonia to see if this technique can differentiate them.

Study Population:

We intend to do an internal pilot study of 6 patients with organic dystonia, 6 patients with clinically definite psychogenic dystonia and 6 age-matched healthy volunteers. We will then perform an analysis to see how many subjects we need to prove or disprove a difference between groups.

Design:

Subjects will have a baseline screening visit, electromyography (EMG) and nerve stimulation, sensory threshold testing, and measurements of brain excitability using motor evoked potentials (MEPs) from transcranial magnetic stimulation (TMS). They will then undergo rapid TMS repetitively paired with stimulation of a nerve in the arm. Outcome variables will again be measured immediately after (T0), 30 minutes (T30) after, and 60 minutes (T60) after the end of brain stimulation.

Outcome Measures

Primary outcome variable: Change in MEP amplitudes at T30 from baseline

Secondary outcome variables:

* Input-output curve parameters (measured at baseline, T0, T30, and T60)
* Temporal discrimination threshold (TDT)

Exploratory Measures

* Short interval intracortical inhibition (SICI), a measure of inhibition in the motor cortex
* Influence of Val66Met BDNF polymorphism on the output variables

Repeated measures analyses of variance (ANOVA) will be used to investigate the following three factors on the outcome variables: time (four levels: baseline, T0, T30 and T60) and muscle (two levels: APB and FDI) as within-subject factor and group (three levels: organic dystonia, psychogenic dystonia, and healthy controls) as between-subjects factor. The model of repeated measures ANOVA will include the interactions between the three factors. If the interaction between muscle and group is significant, the interaction between time and group will be evaluated for each muscle separately. If significance is found for time and/or group, then the evaluation will be followed by Tukey Kramer multiple pair-wise comparisons.

ELIGIBILITY:
* INCLUSION CRITERIA:
* For the organic dystonia group: Primary focal dystonia diagnosed or confirmed by a movement disorders neurologist, confirmed at the initial visit by a study investigator.
* For the psychogenic dystonia group: Clinically established psychogenic dystonia or probable psychogenic dystonia, according to the Fahn and Williams criteria confirmed by a movement disorders neurologist.
* For the healthy volunteers group: Age-matched healthy volunteers three will be age matched to pyschogenic dystonia group, and three will be age matched to organic dystonia group.
* Adult patients (at least18 years old).
* Right handed.
* Ability to provide own consent

EXCLUSION CRITERIA:

* Dystonia affecting the right APB and/or FDI, or inability of the subject to perform full range-of-motion exercises with the right FDI and/or APB.
* Medical condition impairing the subject's ability to comply with the study protocol as judged by study investigator, such as but not limited to seizures, brain tumor, stroke, bipolar disorder, depression, hearing problem, uncontrolled systemic hypertension with values above 170/100, heart disease or lung disease, active respiratory disease needing intervention; and pain preventing lying still for up to 40 minutes.
* Current or prior use of botulinum toxin within 3 months prior to TMS intervention.
* Current or prior use of CNS drugs (including antidepressants, anxiolytics, anticonvulsants, antipsychotics, anti-parkinsonian drugs, hypnotics, stimulants, and/or antihistamines) within 1 week prior to TMS intervention.
* Active drug or alcohol intake more than 7 alcohol drinks/week for women and more than 14 alcoholic drinks/week for men.
* Current pregnancy and lactating women. Menopausal status will be determined by the CNS IRB criteria. In women of childbearing potential, a pregnancy test will be performed at least 24 hours prior to TMS procedures.
* Presence of implanted devices such as pacemakers, medication pumps or defibrillators, metal in the cranium except mouth, history of shrapnel injury or any other condition/device that may be contraindicated
* Inability or unwillingness of subject to provide written informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-06-18; Primary Completion 2016-08-02 (Actual); Study Completion 2016-08-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the motor evoked potential (MEP) amplitude at S50 after 30 minutes from rPAS (T30). | 30 minutes from rPAS

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Avanzino L, Martino D, van de Warrenburg BP, Schneider SA, Abbruzzese G, Defazio G, Schrag A, Bhatia KP, Rothwell JC. Cortical excitability is abnormal in patients with the "fixed dystonia" syndrome. Mov Disord. 2008 Apr 15;23(5):646-52. doi: 10.1002/mds.21801. PMID 18175341
- [Background] Awiszus F. TMS and threshold hunting. Suppl Clin Neurophysiol. 2003;56:13-23. doi: 10.1016/s1567-424x(09)70205-3. No abstract available. PMID 14677378
- [Background] Cheeran B, Talelli P, Mori F, Koch G, Suppa A, Edwards M, Houlden H, Bhatia K, Greenwood R, Rothwell JC. A common polymorphism in the brain-derived neurotrophic factor gene (BDNF) modulates human cortical plasticity and the response to rTMS. J Physiol. 2008 Dec 1;586(23):5717-25. doi: 10.1113/jphysiol.2008.159905. Epub 2008 Oct 9. PMID 18845611